CLINICAL TRIAL: NCT04597619
Title: Evaluation of a Nonopioid Recovery Pathway After Percutaneous Nephrolithotomy
Brief Title: Evaluation of a Nonopioid Recovery Pathway Following Surgery for Kidney Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Rhode Island Hospital (Other); Brown Physicians, Inc. (Other)
Responsible Party: Principal Investigator, David Sobel, M.D., Assistant Professor of Urology, The Miriam Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1574642; P20GM125507 (NIH)
Record Dates: First submitted 2020-10-09; First posted 2020-10-22 (Actual); Results first posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-08

CONDITIONS: Nephrolithiasis
Keywords: Kidney Calculi; Surgery; Nephrolithotomy, Percutaneous
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Pragmatic Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Implementation Cohort (No Intervention): Cohort undergoing PCNL prior to implementation of the novel nonopioid pathway
- Implementation Cohort (Experimental): Cohort undergoing PCNL with implementation of the novel nonopioid pathway
  Interventions: Other: Novel Nonopioid Pathway

INTERVENTIONS:
Other: Novel Nonopioid Pathway — The novel nonopioid pathway consists of preoperative counseling, postoperative standardized orders and standard of care adjunctive and analgesic medications, specialized discharge instructions and written patient instructions regarding medications and activity.
  Arms: Implementation Cohort

SUMMARY:
Evaluation of a nonopioid recovery pathway after percutaneous nephrolithotomy is a pragmatic pilot study that will apply the knowledge and experience gained with development of an outpatient opioid reduction protocol to percutaneous nephrolithotomy (PCNL). We have previously demonstrated that outpatient ureteroscopy and stent placement without postoperative opioid prescriptions is possible in the vast majority of patients. The success of this is dependent upon a multimodal approach to the patient's experience of undergoing endoscopic kidney stone surgery (ureteroscopy) and focuses on the preoperative, perioperative, and postoperative stages of intervention. Our hypothesis is that a novel nonopioid pathway after PCNL is both feasible and safe and will reduce postoperative prescriptions for opioids without impacting clinical outcomes, patient satisfaction or outpatient resources.

DETAILED DESCRIPTION:
Evaluation of a nonopioid recovery pathway after percutaneous nephrolithotomy is a pragmatic pilot study which will prospectively compare a cohort undergoing PCNL prior to implementation of the novel nonopioid pathway undergoing the same procedure utilizing the novel nonopioid pathway. Current standard of care following PCNL remains the routine prescription of opioid medications for pain control.

Evaluation of a nonopioid recovery pathway after percutaneous nephrolithotomy has three specific aims:

1. Demonstrate feasibility and acceptability of the novel nonopioid protocol and describe the barriers to enrollment and reasons for drop out. The feasibility of the protocol will be measured by dropout of enrolled patients and the acceptability of protocol will be measured by number of enrolled patients / patients approached and patient satisfaction via a validated questionnaire.
2. Describe what adverse events occur to those on the nonopioid protocol as compared to the standard of care. Adverse events occurring as an inpatient will be measured by nursing and physician reporting, and as an outpatient via patient self-reporting, electronic medical records of emergency department visits and telephone calls to clinic.
3. Begin to reduce overall opioid prescription writing for patients undergoing PCNL at the academic institution. The electronic medical records will be queried for prescriptions written at discharge. The state Opioid Prescription Monitoring Program (PMP) will be queried for a 30-day period following surgery.

After written consent and enrollment, patients will undergo preoperative counseling regarding pain after PCNL in the preoperative holding area prior to surgery. The patient will then undergo percutaneous nephrolithotomy. No procedural changes will be made for study participants. Postoperatively, patients will be admitted to the post-anesthesia care unit and standard of care adjunctive and analgesic medications will be administered. The patient will be admitted to the floor following surgery and postoperative specialized nonopioid PCNL pathway orders will be communicated to nursing staff. The patient's pain will be treated with multimodal nonopioid analgesic agents. Opioid medications will not be withheld for patients with severe pain. On postoperative day one, the patient will be assessed for discharge as in standard of care. They will be asked about their perceived need for a prescription for opioids. If requested, the patient will be given a prescription for a limited quantity of opioids. Nursing staff will complete specialized discharge instructions and patients will be given written instructions regarding medications and activity. Patients will be seen in 7-10 days for stent removal in the office per standard of care, and will complete a validated quality of life survey for pain after kidney stone surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary percutaneous nephrolithotomy at a single academic hospital site.

Exclusion Criteria:

* Patients will be excluded if currently taking opioids for chronic pain, undergoing concurrent non-PCNL procedure, second-look PCNL (subsequent PCNL after primary PCNL), or present with Chronic Kidney Disease Stage >3 or glomerular filtration rate < 50 mL/min/1.73m2 at time of surgery.
* Patients with allergy to NSAIDs or have history of NSAID related GI bleeding or ulcers will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-06-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sobel D, Caffery P, James E, Ortiz R, Peat A, Tucci C, Pareek G. A prospective study to determine the safety and feasibility of opioid-free discharge after percutaneous nephrolithotomy. Transl Androl Urol. 2025 May 30;14(5):1379-1390. doi: 10.21037/tau-2024-692. Epub 2025 May 27. PMID 40529026

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-Implementation Cohort: Cohort undergoing percutaneous nephrolithotomy (PCNL) prior to implementation of the novel nonopioid pathway
- Implementation Cohort: Cohort undergoing percutaneous nephrolithotomy (PCNL) with implementation of the novel nonopioid pathway
  Novel Nonopioid Pathway: The novel nonopioid pathway consists of preoperative counseling, postoperative standardized orders and standard of care adjunctive and analgesic medications, specialized discharge instructions and written patient instructions regarding medications and activity.
Period: Overall Study
Arm/Group | Pre-Implementation Cohort | Implementation Cohort
Started | 20 | 10
Completed | 14 | 6
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Implementation Cohort | Implementation Cohort | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 4 | 14
  >=65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 10 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 5 | 17
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Previous nephrolithiasis requiring surgery [Count of Participants; unit: Participants] | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Protocol Feasibility
Description: Number of enrolled patients / patients approached
Time Frame: 1 year or until subject accrual is complete
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort | Implementation Cohort
Number analyzed (Participants) | 20 | 10
Participants | 14 | 10

2. Primary Outcome: Adherence to the Protocol
Description: Dropout of enrolled patients
Time Frame: 30 days after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort | Implementation Cohort
Number analyzed (Participants) | 14 | 10
Participants | 14 | 6

3. Primary Outcome: Adverse Events
Description: Adverse events (AEs) while inpatient and following discharge
Time Frame: Day of procedure to 30 days after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort | Implementation Cohort
Number analyzed (Participants) | 14 | 6
Participants | 0 | 0

4. Primary Outcome: Opioid Free Discharge
Description: Whether subject is discharged with prescription for opioids or not
Time Frame: Within 24 hours of discharge from hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort | Implementation Cohort
Number analyzed (Participants) | 14 | 6
Participants | 10 | 6

5. Secondary Outcome: Postoperative Inpatient Opioid Utilization
Description: Postoperative inpatient intravenous opioid utilization (morphine milliEquivalents / kg / day)
Time Frame: 24-48 hours
Measure: Median (Inter-Quartile Range); unit: morphine mEq / kg / day
Arm/Group | Pre-Implementation Cohort | Implementation Cohort
Number analyzed (Participants) | 14 | 6
morphine mEq / kg / day | 4.0 [2.0 to 4.0] | 0 [0 to 0]

6. Secondary Outcome: Discharge Opioid Prescriptions
Description: Opioid prescriptions written at time of discharge (morphine milliEquivalents / kg / day)
Time Frame: At time of discharge, average of postoperative day 1
Measure: Median (Inter-Quartile Range); unit: morphine mEq / kg / day
Arm/Group | Pre-Implementation Cohort | Implementation Cohort
Number analyzed (Participants) | 14 | 6
morphine mEq / kg / day | 30.0 [20.0 to 30.0] | 0 [0 to 0]

7. Secondary Outcome: Nonopioid Discharge Medications
Description: Nonopioid medications given for pain
Time Frame: At time of discharge, average of postoperative day 1
Reporting Status: Not Posted

8. Secondary Outcome: Length of Stay (Hours)
Description: Length of inpatient stay (hours)
Time Frame: 24-48 hours
Measure: Median (Inter-Quartile Range); unit: day(s)
Arm/Group | Pre-Implementation Cohort | Implementation Cohort
Number analyzed (Participants) | 14 | 6
day(s) | 1 [1 to 1] | 1 [1 to 1]

9. Secondary Outcome: Clinic Calls
Description: Quantitative number of telephone calls to clinic for pain / discomfort within 30 days via documentation in electronic medical record
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort | Implementation Cohort
Number analyzed (Participants) | 14 | 6
Participants | 1 | 1

10. Secondary Outcome: Refill Requests
Description: Quantitative number of requests for refills of opioid prescriptions within 30 days via documentation in EMR
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort | Implementation Cohort
Number analyzed (Participants) | 14 | 6
Participants | 0 | 0

11. Secondary Outcome: Emergency Department Visits
Description: Quantitative number of subject presentations to emergency department for pain within 30 days via documentation in EMR
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort | Implementation Cohort
Number analyzed (Participants) | 14 | 6
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Day of subject's surgery to thirty (30) days following stent removal.
Arm/Group | Pre-Implementation Cohort | Implementation Cohort
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6
Other Adverse Events (participants affected / at risk) | 0/14 | 0/6

LIMITATIONS AND CAVEATS:
Small pragmatic pre- and post- study without randomization designed to evaluate feasibility and safety only. Enrollment/accrual hampered by COVID-19 pandemic where healthcare rationing and other emergency response protocols limited screened patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT04597619/Prot_SAP_000.pdf